CLINICAL TRIAL: NCT05606523
Title: Can Fecal Microbiota Transplantation of Cachectic Patients with Pancreas Cancer Impair Body Weight Gain in Germ-free Mice? the EXTRA Study
Brief Title: Microbiota and Pancreatic Cancer Cachexia
Acronym: EXTRA
Status: Recruiting | Type: Observational
Sponsor: Genton Graf Laurence (Other)
Responsible Party: Sponsor-Investigator, Genton Graf Laurence, Principal Investigator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: 2022-00820
Record Dates: First submitted 2022-08-25; First posted 2022-11-04 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Pancreatic Cancer; Microbiota; Cachexia
MeSH Terms: conditions — Pancreatic Neoplasms; Cachexia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — feces, saliva, blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Cachectic patients with pancreatic cancer: Measurements and sample collection at one timepoint.
- Non-cachectic patients with pancreatic cancer: Measurements and sample collection at one timepoint.
- Healthy volunteers: Measurements and sample collection at one timepoint.

SUMMARY:
This monocentric study aims at evaluating the effects of fecal microbiota transplantation from newly diagnosed cachectic and non-cachectic pancreatic cancer patients, and healthy volunteers on several cachexia-related parameters of germ-free mice.

DETAILED DESCRIPTION:
Aim: Evaluating the effects of fecal microbiota transplantation (FMT) from 6 newly diagnosed cachectic and 6 non-cachectic pancreatic cancer patients, and 12 healthy age-and sex-matched volunteers on several cachexia-related parameters of 96 germ-free mice (4 per donor) over a 30-day period. The fecal material of all 12 pancreatic cancer patients will be collected at diagnosis before any cancer treatment onset.

Hypothesis: FMT of cachectic patients with pancreas cancer, naïve of any anti-cancer treatment and artificial nutrition, into germ-free mice impairs weight gain, in contrast to FMT of non-cachectic patients and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

Patients with pancreatic cancer (n=12)

* ≥18 years and
* Newly diagnosed of pancreatic adenocarcinoma (local or metastatic) and
* Tube feeding or parenteral nutrition ≤ 14 days

Cachectic pancreatic cancer patients (n=6)

* Cachexia according to the Fearon criteria 1: involuntary weight loss >5% over the last 6 months, or any level of weight loss >2% and a BMI <20 kg/m2 or sarcopenia. Sarcopenia will be diagnosed by BIA (fat-free mass index is <17 kg/m2 in men and <15 kg/m2 in women) 81, and not by CT, as it is faster and can be performed at the bedside of the patient. Non-cachectic pancreatic cancer patients (n=6)
* Normal nutritional state: weight stability (± 2% of habitual weight) over the last 6 months, no anorexia before the diagnosis (appetite rating on a visual analogue scale of 100mm), no known impaired glucose tolerance.

Healthy matched subjects (n=12)

* ≥18 years and
* BMI between 18.5 and 30 kg/m2 and
* Absence of chronic or acute disease and
* Matching for gender and age (± 5 years) with an included pancreatic cancer patient

Exclusion Criteria:

* < 18 years or
* Inability to give consent or
* Insufficient knowledge of project language (French, German) or
* Pancreatic adenocarcinoma already treated by chemo- or radiotherapy, or major surgery as duodenopancreatectomy or biliary diversion
* Known rheumatologic or immunologic diseases
* Therapeutic antibiotics or immunosuppressive drugs (for instance glucocorticoids, cytostatics, antibodies) in the 30 days preceding the inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will consider the fecal samples of 12 patients at diagnosis of pancreatic cancer including 6 patients with cachexia and 6 patients without cachexia, and therefore naïve of any anti-cancer treatment and artificial nutritional support. We will also include 12 healthy volunteers matched for gender and age (± 5 years) with the pancreatic cancer patients.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Body weight changes in mice after fecal material transplantation. | Between days 0 and 30
  Body weight (g)

SECONDARY OUTCOMES:
Differences in fecal microbiota | at diagnosis
  by 16S rRNA gene amplicon sequencing and functional profiles by metagenomic sequencing between cachectic patients non-cachectic patients and healthy volunteers
Body weight | at diagnosis
  in kilograms between cachectic patients non-cachectic patients and healthy volunteers
Waist-to-hip ratio | at diagnosis
  waist circumference (cm) and hip circumference (cm) between cachectic patients non-cachectic patients and healthy volunteers
Fat mass | at diagnosis
  by bioelectrical impedance analysis (BIA) between cachectic patients non-cachectic patients and healthy volunteers
Fat-free mass | at diagnosis
  by bioelectrical impedance analysis (BIA) between cachectic patients non-cachectic patients and healthy volunteers
Muscle mass | at diagnosis
  surfaces of the paraspinal and abdominal wall muscles at the level of L3-L4 disk space by CT for pancreatic cancer patients
Nutritional intake | at diagnosis
  by 3-day food diary between cachectic patients non-cachectic patients and healthy volunteers
Resting energy expenditure (REE) | at diagnosis
  by indirect calorimetry between cachectic patients non-cachectic patients and healthy volunteers
Appetite | at diagnosis
  by visual analogue scale ranging from 0 to 100 mm between cachectic patients non-cachectic patients and healthy volunteers
Appetite | at diagnosis
  by fasting level of plasma ghrelin between cachectic patients non-cachectic patients and healthy volunteers
Appetite | at diagnosis
  by fasting level of plasma leptin between cachectic patients non-cachectic patients and healthy volunteers
Appetite | at diagnosis
  by fasting level of plasma glucagon-like peptide-1 (GLP-1) between cachectic patients non-cachectic patients and healthy volunteers
Appetite | at diagnosis
  by fasting level of plasma neuropeptide Y between cachectic patients non-cachectic patients and healthy volunteers
Appetite | at diagnosis
  by fasting level of plasma cholecystokinin between cachectic patients non-cachectic patients and healthy volunteers
Homeostatic model assessment (HOMA)-score | at diagnosis
  by fasting glycemia (mmol/l) and fasting insulinemia (mU/ml)) between cachectic patients non-cachectic patients and healthy volunteers
Glycemia | at diagnosis
  by fasting glycemia (mmol/l) between cachectic patients non-cachectic patients and healthy volunteers
Insulinemia | at diagnosis
  by fasting insulinemia (mU/ml) between cachectic patients non-cachectic patients and healthy volunteers
Physical function | at diagnosis
  by handgrip strength between cachectic patients non-cachectic patients and healthy volunteers
Physical activity | at diagnosis
  by the International Physical Activity Questionnaire (IPAQ) between cachectic patients non-cachectic patients and healthy volunteers
Quality of life | at diagnosis
  by the European Organisation for Research and Treatment of Cancer questionnaire (EORTC QLQ-C30) between cachectic patients non-cachectic patients and healthy volunteers
Mortality | at diagnosis
  by tumor progression between cachectic patients non-cachectic patients
Oral microbiota | at diagnosis
  by 16SrRNA gene amplicon sequencing and metagenomic sequencing between cachectic patients non-cachectic patients and healthy volunteers
Epithelial permeability | at diagnosis
  by fasting levels of plasma zonulin between cachectic patients non-cachectic patients and healthy volunteers
Epithelial permeability | at diagnosis
  by fasting levels of plasma lipopolysaccharide-binding protein between cachectic patients non-cachectic patients and healthy volunteers
Epithelial permeability | at diagnosis
  by fasting levels of plasma glucagon-like peptide-2 between cachectic patients non-cachectic patients and healthy volunteers
GALT function and systemic inflammation | at diagnosis
  by fasting plasma level of C-reactive protein (CRP) and cytokines between cachectic patients non-cachectic patients and healthy volunteers
GALT function and systemic inflammation | at diagnosis
  by peripheral blood T regulatory cells (Tregs) levels and phenotype between cachectic patients non-cachectic patients and healthy volunteers
GALT function and systemic inflammation | at diagnosis
  by myeloid derived suppressor cells (MDSC) levels and phenotype between cachectic patients non-cachectic patients and healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Genton Graf, Prof, Principal Investigator — Geneva University Hospitals (HUG)
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland